CLINICAL TRIAL: NCT02947061
Title: S1 Plus Docetaxel Versus Capecitabine Plus Docetaxel First-line Treatment in Patients With Advanced Breast Cancer: a Phase 2, Prospective,Multicenter, Randomised Study
Brief Title: S1 Plus Docetaxel Versus Capecitabine Plus Docetaxel First-line Treatment in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, Professor and Director, Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-033
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer Recurrent
Keywords: Advanced Breast Cancer,first treatment, S1, Capecitabine
MeSH Terms: interventions — S 1 (combination); Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- test group (Experimental): S1 plus Docetaxel ：S-1 80mg to 120 mg per day on Days 1-14, every 21 days; Docetaxel 75mg/m2 on Day 1
  Interventions: Drug: S1 plus Docetaxel
- control group (Active Comparator): Capecitabine plus Docetaxel ：Capecitabine 1,000 mg/m2 per day on Days 1-14, every 21 days; Docetaxel 75mg/m2 on Day 1
  Interventions: Drug: Capecitabine plus Docetaxel

INTERVENTIONS:
Drug: S1 plus Docetaxel — S1 80mg to 120 mg per day on Days 1-14, every 21 days; Docetaxel 75mg/m2 on Day 1
  Arms: test group
Drug: Capecitabine plus Docetaxel — Capecitabine 1,000 mg/m2 per day on Days 1-14, every 21 days; Docetaxel 75mg/m2 on Day 1
  Arms: control group

SUMMARY:
To compare the progression free survival(PFS) and safety of TS-S vs. TX-X in Patients With Advanced Breast Cancer first-line treatment

DETAILED DESCRIPTION:
To compare progression free survival (PFS) of the S-1 combined with docetaxel followed by maintenance treatment with S-1 and capecitabine combined with docetaxel followed by maintenance therapy with capecitabine in patients with advanced breast cancer first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 75;
* ECOG 0-2, The expected survival time more than 3 months;
* Histologically or cytologically proven locally advanced or advanced HER-2 negative breast cancer;
* No chemical treatment after Cancer recurrence;
* At least one measurable disease ( as per RECIST1.1);
* Adequate bone marrow functions (ANC ≥1.5×109 /L, PLT ≥100×109 /L, HB ≥90 g/L);
* Adequate renal functions(serum creatinine ≤ 1.5 ULN; creatinine clearance≥50 ml/min);
* liver functions (serum bilirubin ≤ 1.5ULN, AST/ALT ≤ 2.5 ULN);
* Written informed consent;
* Pregnancy test (serum or urine) within 7 days of entry and willing to use the appropriate method of contraception.

Exclusion Criteria:

* Previously chemotherapy with cytotoxic drugs
* Pregnant, lactating women Did not take effective contraceptive measures
* Adjuvant chemotherapy/ neoadjuvant chemotherapy with 5-FU-based chemotherapy or Paclitaxel -based chemotherapy within 1 year after recurrence;
* Her-2 positive or unknown
* Other trails Before 4weeks
* Affection of the absorption of drugs(Unable to swallow、after gastrectomy、Chronic diarrhea and intestinal obstruction
* Organs with rapid progression of invasion(Liver and lung lesions more than 1/2 organ area or hepatic insufficiency)
* Central nervous system disorders or mental disorders
* For docetaxel or fluorouracil or Twain 80 had serious adverse reactions or Allergy to 5-FU
* Severe upper gastrointestinal ulcer or absorption dysfunction syndrome
* Abnormal blood routine (ANC <1.5×109 /L, PLT <100×109 /L, HB <90 g/L);
* Renal functions(serum creatinine > 1.5 ULN);
* Liver functions (serum bilirubin > 1.5ULN
* Brain metastases out of control
* Other unapplicable

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 years

SECONDARY OUTCOMES:
overall survival | 1 year
objective response rate | 2 years
Disease control rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, M.D., Principal Investigator — Chinese Academy of Medical Sciences; Guohui Han, M.D., Principal Investigator — Tumor Hospital of Shanxi Province
Locations (1):
- No.17 panjiayuannanli, Chaoyang District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No